CLINICAL TRIAL: NCT06307535
Title: Meaning-Centered Psychotherapy to Meet Palliative Care Needs of Cancer Caregivers
Brief Title: A Study of Meaning-Centered Psychotherapy for Caregivers to People With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Allison Applebaum, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-24-01356
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Caregiver Burden; Caregiver Burnout; Caregiver Stress Syndrome
Keywords: Caregiver; Caregiver Stress Syndrome; Caregiver Burden; Caregiver Burnout; Meaning-Centered Psychotherapy; 23-376
MeSH Terms: conditions — Caregiver Burden | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meaning-Centered Psychotherapy for Caregivers (Experimental): Meaning-Centered Psychotherapy for Caregivers/MCP-C
  Interventions: Behavioral: Meaning-Centered Psychotherapy for Caregivers
- Supportive Psychotherapy for Caregivers (Active Comparator): Supportive Psychotherapy for Caregivers/SP-C standard of care
  Interventions: Behavioral: Supportive Psychotherapy for Caregivers

INTERVENTIONS:
Behavioral: Meaning-Centered Psychotherapy for Caregivers — MCP-C is a stakeholder-informed, innovative, manualized intervention designed to assist caregivers to connect to a sense of meaning and purpose in life, despite the challenges of caregiving.
  Other Names: MCP-C
  Arms: Meaning-Centered Psychotherapy for Caregivers
Behavioral: Supportive Psychotherapy for Caregivers — Standard of care supportive psychotherapy
  Other Names: SP-C
  Arms: Supportive Psychotherapy for Caregivers

SUMMARY:
Participants will complete 1 set of questionnaires about 2 weeks before beginning their Meaning-Centered Psychotherapy for Caregivers/MCP-C or standard Supportive Psychotherapy for Caregivers/SP-C sessions. These questionnaires will ask about participants' sense of meaning and purpose in life, spiritual well-being, depression and/or anxiety, and social support. Participants will then be assigned to receive either MCP-C or SP-C for 7 sessions. Participants will complete additional sets of questionnaires about 2 weeks, 6 months, and 12 months after their last session of MCP-C or SP-C. It will take between 35 and 50 minutes to complete each set of questionnaires.

After participants complete the MCP-C or SP-C sessions and all 4 sets of questionnaires, their participation in this study will end. If participants decide not to complete all 7 sessions, they may still choose to complete the questionnaires.

Participants may remain in the study and continue to receive all 7 sessions of MCP-C or SP-C even if their loved one passes away.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over;
* As per self-report, a current caregiver to a patient with Stage III or IV solid tumor cancer currently receiving medical care of any kind (e.g., curative, palliative);
* Experiences distress as evidenced by a score of 4 or greater on the Distress Thermometer (DT) and an indication that this distress is associated with caregiving;
* As per self-report, can read and understand English;
* As per self-report, residing in New York, New Jersey, or Florida, or have the ability to complete sessions while complying with current telehealth regulations.

Exclusion Criteria:

* Participant does not have a reasonable understanding of the study activities by the judgment of the consenting professional;
* Engagement in regular individual psychotherapeutic support that the participant is unable or unwilling to put on hold for the course of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved primary outcomes | Up to 1 year
  Evaluate the efficacy of MCP-C versus SP-C in improving primary outcomes (i.e., sense of meaning in life, spiritual well-being) immediately post-treatment and explore maintenance in gains up to 1 year.
Life Attitude Profile-Revised (LAP-R) | Up to 1 year
  Life Attitude Profile-Revised (LAP-R) - used to measure sense of meaning in life.
  The LAP-R is a 48-item instrument. Each item is rated on a 7-point Likert scale ranging from "strongly agree" to "strongly disagree." Full scale ranges from 30 to 210 with a higher score indicating a greater sense of meaning in life and a more positive attitude towards life.
FACIT Spiritual Well-Being Scale (SWBS) | Up to 1 year
  The Spiritual Well-Being Scale (SWBS) - used to measure spiritual well-being.
  The SWBS is a 12-item instrument. Each item is scored from 1 to 5. Negatively worded items are reverse scored. The measure generates two sub-scales: Faith/Spirituality (0-16) and Meaning/Peace (0-32). Full scale ranges from 0 to 48. Higher scores indicate a greater sense of spiritual well-being.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Up to 1 year
  Hospital Anxiety and Depression Scale (HADS) - measures anxiety and depression.
  14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating poorer health outcome.
Benefit Finding Scale (BFS) | Up to 1 year
  Benefit Finding Scale (BFS) - measures benefit finding.
  The BFS is a 17-item instrument. Each item is scored from 1-5 (not at all, a little bit, somewhat, quite a bit, or very much). Full scale ranges from 17 to 85, with higher scores indicating greater benefit finding.
Caregiver Reaction Assessment (CRA) | Up to 1 year
  Caregiver Reaction Assessment (CRA) - measures caregiver burden.
  The CRA is a 24-item instrument. Full scale ranges from 24 to 120, with higher scores indicating greater caregiving burden
Duke-UNC Functional Social Support Questionnaire (FSSQ) | Up to 1 year
  Duke-UNC Functional Social Support Questionnaire (FSSQ) - measures social support.
  The FSSQ is an 8-item instrument. Each item is scored on a scale of 5-1 where 5=as much as I would like; 4=almost as much as I would like; 3=some, but would like more; 2=less than i would like, and 1=much less than I would like. Full scale ranges from 0 to 44 with higher scores indicating a higher degree of satisfaction related to social support.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, FAPOS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (8):
- United States (8):
  - University of Miami (Data Collection AND Data Analysis), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Requests for deidentified individual participant data can be made from the date of publication until six years post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: MSIPinfo@mssm.edu
Time Frame: Until six years post publication
URL: https://ip.mountsinai.org/contact-msip/